CLINICAL TRIAL: NCT02718573
Title: Impact of Interferon-free Treatment for Hepatitis C Virus (HCV) on Blood Cells and Factors in Blood
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Andrea Branch, Andrea D. Branch PhD, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 14-2222
Record Dates: First submitted 2016-03-18; First posted 2016-03-24 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Hepatitis C; HCV; Liver Transplant
Keywords: Hepatitis C; Interferon-free; DDA's
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-liver transplants with HCV
- Liver transplants with HCV

SUMMARY:
The objectives of the study are to determine the impact of interferon-free treatment for the hepatitis C virus (HCV) on peripheral blood immune cell phenotype and soluble immune-related proteins in blood, while controlling for genetic polymorphisms known to impact HCV-related immune responses, and to determine the impact of the therapy on the emergence of drug-resistant HCV. The study design is informed by the researchers recent investigations of patients receiving HCV treatment. About 4% of patients who had not undergone liver transplantation experienced hepatic decompensating or another serious event. There were several cases of bacterial infection and two cases with elevated markers of autoimmune processes. These events suggest that treatment altered immune responses. About 25% of patients who had undergone liver transplantation experienced hepatic decompensating or another serious adverse event. The long term goal is to understand the pathophysiology of these complications and determine whether HCV treatment can cause an immune reconstitution syndrome in susceptible patients, while improving antimicrobial defenses in others

DETAILED DESCRIPTION:
The objectives of the study are to determine the impact of interferon-free treatment for the hepatitis C virus (HCV) on peripheral blood immune cell phenotype and soluble immune-related proteins in blood, while controlling for genetic polymorphisms known to impact HCV-related immune responses, and to determine the impact of the therapy on the emergence of drug-resistant HCV. The study design is informed by the researchers' recent investigations of patients receiving HCV treatment. About 4% of patients who had not undergone liver transplantation experienced hepatic decompensation or another serious event. There were several cases of bacterial infection and two cases with elevated markers of autoimmune processes. These events suggest that treatment altered immune responses. About 25% of patients who had undergone liver transplantation experienced hepatic decompensation or another serious adverse event. The long term goal is to understand the pathophysiology of these complications and determine whether HCV treatment can cause an immune reconstitution syndrome in susceptible patients, while improving antimicrobial defenses in others The main questions/objectives to be addressed are (1) to determine the effect of HCV treatment on the profile of immune cells in blood as assessed by cytometry time of flight (CyTOF) multiparameter analysis, while controlling for genetic polymorphisms known to be associated with HCV-related immune responses and, (2) to determine the effect of treatment on factors/proteins in blood that may be related to immunity and inflammation.

Background: New treatments for HCV are significantly more effective than past treatments. They utilize direct acting antiviral drugs (DAA) and many do not include interferon. The goal of treatment is to achieve a sustained virological response (SVR). An SVR is indicated by the absence of detectable HCV RNA in blood 12 weeks after the end of treatment (EOT); this is called SVR12. The researchers recently investigated outcomes of 514 non-liver transplant (LT) patients and 43 LT patients who initiated treatment between Dec 2013 and June 2014. Several patients developed increased levels of markers of autoimmune processes and/or experienced a bacterial infection. Investigators at other institutions recently reported evidence that DAA treatment enhances immune cell activation. The combination of the investigators' observations and the observations of others indicates that a detailed investigation is needed to understand the events leading to increased immune cell activity and to determine the factors that may increase the risk of serious adverse events.

ELIGIBILITY:
Inclusion for non-LT patients:

* Adult
* Not pregnant
* Positive test for HCV RNA and planning to start interferon-free treatment soon
* Not HIV infected
* Able and willing to travel to Mount Sinai at the time points need for blood draws--prior to the start of treatment (within one month of the actual start date), at the 4th week of treatments (plus or minus two weeks), at the 12th week of treatment (plus or minus two weeks).
* Must understand and speak English
* Medically stable
* Willing to sign informed consent and participate

Inclusion criteria for LT patients:

* All of the above
* At least 6 months post-LT
* On stable immunosuppressive medications for at least 3 months LT only (no other organ transplant, such as kidney)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified by their health care providers, including the co-investigators, who will describe the study to potential participants and inform the research team of patients who are interested in participating.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
cytometry time of flight (CyTOF) | up to week 14
  the profile of immune cells in blood as assessed by cytometry time of flight (CyTOF) multiparameter analysis

SECONDARY OUTCOMES:
CD8 T cells | Baseline and week 14
  Change in the percentage of CD8 Tcells level
HCV resistance mutations | up to week 14
  Incidence of emergence of HCV resistance mutations

CONTACTS AND LOCATIONS:
Overall Officials: Andrea D. Branch, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes